CLINICAL TRIAL: NCT06010992
Title: A Clinical Study Evaluating the Potential Benefit of Nitazoxanide in Patients With Type 2 Diabetes Mellitus
Brief Title: Nitazoxanide as Adjuvant Therapy in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Principal Investigator, Eman Ghonaim, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MD53/3/23
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — nitazoxanide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): 35 Patients with type 2 diabetes receiving treatment with metformin and dipeptidyl peptidase-4 (DPP-4) inhibitors (such as vildagliptin).
- Group 2 (Experimental): 35 Patients with type 2 diabetes receiving nitazoxanide 500 mg orally twice daily in addition to metformin and dipeptidyl peptidase-4 (DPP-4) inhibitors (such as vildagliptin).
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide oral capsules 500 mg twice daily
  Arms: Group 2

SUMMARY:
Diabetes mellitus (DM) is a complex metabolic disorder characterized by hyperglycemia and abnormalities in carbohydrate, fat, and protein metabolism. Despite the advancement in anti-diabetic drug therapy, most patients fail to achieve optimal glycemic control. This highlights the need for more effective strategies to control type 2 diabetes mellitus.

Nitazoxanide (NTZ), a broad-spectrum anti-infective drug with activity against various protozoa, helminthes, bacteria, and viruses, was identified as peroxisome proliferative activated receptor gamma (PPARγ) agonist using one dimensional drug profile matching. Additionally, it improved insulin sensitivity in insulin-resistant type 2 diabetic rats. Therefore, this study is designed to evaluate the efficacy of nitazoxanide as adjunctive therapy in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Glycated hemoglobin (HbA1c) between 7% and 9%.
* Body mass index ≥ 25 kg/m2

Exclusion Criteria:

* Pregnant or nursing women.
* Type 1 diabetes mellitus.
* Liver disease (alanine aminotransferase > 3 upper normal limit).
* Kidney disease (estimated glomerular filtration rate < 60 ml/min/1.73 m2).
* Inflammatory bowel diseases.
* History of allergy and/or adverse reactions to the drugs used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | 12 weeks
  Fasting blood glucose and glycated hemoglobin

SECONDARY OUTCOMES:
Insulin resistance | 12 weeks
  fasting insulin level with HOMA-IR calculation
Lipid profile | 12 weeks
  Serum levels of total cholesterol, LDL, HDL, and triglycerides
Serum levels of A-kinase anchoring protein 1 | 12 weeks
Serum levels of asprosin | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eman Ghonaim, Principal Investigator — Assistant Lecturer, Faculty of Pharmacy, Tanta University
Locations (2):
- Egypt (2):
  - Faculty of medicine, Tanta University, Tanta, El-Gharbia
  - Faculty of Medicine, Menoufia University, Shibīn al Kawm, Menoufia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghonaim EM, Ibrahim OM, Hegazy SK, Farrag WF, Badr HR. Repurposing nitazoxanide in type 2 diabetes mellitus: a randomized controlled trial. Endocrine. 2025 Nov;90(2):596-604. doi: 10.1007/s12020-025-04387-5. Epub 2025 Aug 15. PMID 40815384